CLINICAL TRIAL: NCT02685371
Title: Septal Shift for the Diagnosis of COnstrictive Pericarditis: The Impact of Inspiratory Effort Quantification on Deep Breathing Manoeuvres (SCOPED)
Brief Title: Septal Shift for the Diagnosis of COnstrictive Pericarditis: The Impact of Inspiratory Effort Quantification on Deep Breathing Manoeuvres
Acronym: SCOPED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Paul Farand, M.D., Université de Sherbrooke
Other Study IDs: MP-31-2016-1083
Record Dates: First submitted 2016-01-13; First posted 2016-02-18 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Constrictive Pericarditis
MeSH Terms: conditions — Pericarditis, Constrictive | interventions — Respiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Breathing effort type: Current known criteria for constrictive pericarditis will be test under: 1- spontaneous breathing 2- Breathing with a negative pressure of -15 to - 30 cm of water 3- Breathing with a negative pressure of more than - 30 cm of water.
  Interventions: Behavioral: Breathing

INTERVENTIONS:
Behavioral: Breathing — Subjects will have to breath 1- Spontaneously 2- to produce a negative pressure of -15 to -30 cm of water and 3- to produce a negative pressure more than -30 cm of water.

SUMMARY:
This study will evaluate the effect of deep breathing manoeuvres on inter ventricular interdependency physiology. By providing further insight in this basic physiology we want to add more comprehensive data in favor or not of constrictive pericarditis diagnostic criteria currently used in cardiovascular magnetic resonance.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 80 years old
* Normal transthoracic echocardiogram if older than 41 years old
* Normal standardized history and physical examination
* Normal blood pressure (<130/80)
* Normal 12-lead ECG at rest.

Exclusion Criteria:

* No prior pulmonary or cardiac diseases
* Unexplained symptoms that could be related to a heart or pulmonary problems.
* Symptoms of or active cardiovascular or pulmonary problems
* Hepatic or kidney dysfunction
* Blood cell dyscrasia
* Cardiovascular risk factor (smoking, hypertension, dyslipidemia, diabetes)
* Obesity (BMI > 30)
* Pregnancy or pregnancy in the last year
* Cardiac congenital anomalies discovered during the cardiovascular magnetic resonance
* Current medication with cardiovascular side effects known (diuretics, beta-blockers, calcium channel blockers)
* Contraindication to cardiovascular magnetic resonance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population consists of healthy subjects not know for any cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-02 (Estimated); Study Completion 2020-02

PRIMARY OUTCOMES:
Measurement of the interventricular septum position between inspiration and expiration as assessed by CMR. | Immediate
  Analysis of respiratory-related septal excursion. The relative position of the septum can be obtained by dividing the distance between RV free wall and septum by the biventricular distance. If done during inspiration and expiration, at early ventricular filling, the respiratory-related septal excursion can be quantified.

SECONDARY OUTCOMES:
Presence or absence (categorical variable) of a diastolic bounce as assessed by CMR. | Immediate
  Diastolic bounce corresponds to a displacement of inter ventricular septum towards de left ventricle during the protodiastolic period.
Measurement of the variation of flow through the mitral and tricuspid valve between inspiration and expiration as assessed by CMR. | Immediate
  Real-Time Phase-Contrast acquisition using a custom-made sequence with through-plane velocity encoding to simultaneously measure MV and TV inflow velocities by prescribing a slice position across both atrioventricular valves from a horizontal long-axis view.
Biventricular Index: measurement of the heart contour between inspiration and expiration as assessed by CMR. | Immediate
  Short axis cross section through the mid ventricle. The epicardial tracings is performed in end expiration and end inspiration. The end inspiratory epicardial tracing is divided by the end expiratory epicardial tracing to obtain the biventricular index
Presence or absence (categorical variable) of diastolic flow reversal in inferior vein cave as assessed by cardiovascular magnetic resonance (CMR). | Immediate
  Real-time cine imaging of the inferior vein cave for 10 s
Presence or Absence of lack of myocardial slippage in relation to the pericardium as assessed by CMR (tagging sequence) | Immediate
  Four-chamber tagged cardiac magnetic resonance image showing lack of slippage between parietal and visceral pericardia. The tag lines break between parietal and visceral pericardia during the cardiac cycle in a normal heart. In constrictive pericarditis, the tag lines do not break.
Measurement of the relative atrial volume ratio as assessed by CMR. | Immediate.
  The relative atrial volume ratio (RAR) is defined as the left auricular (LA) volume divided by right auricular (RA) volume. For the LA volume, the biplane area- length method will be used. For the RA volume, the monoplane area-length formula will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Paul, Sherbrooke, Quebec, Canada